CLINICAL TRIAL: NCT01451229
Title: An Open-Label, Single-dose Administration Study of the Pharmacokinetics and Pharmacodynamics of Higenamine, Administered Intravenously Injection to Healthy Chinese Subjects
Brief Title: Pharmacokinetics and Pharmacodynamics of Higenamine in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-PK003
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Healthy
Keywords: pharmacokinetics; pharmacodynamics
MeSH Terms: interventions — higenamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: higenamine — infused intravenously with higenamine at the escalating doses from 0.5 ug/kg/min through 1.0 ug/kg/min and 2.0 ug/kg/min to 4.0 ug/kg/min, each dose being given for 3 minutes

SUMMARY:
The purpose of this study is to assess the pharmacokinetics and pharmacodynamics of higenamine in healthy Chinese subjects

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following inclusion criteria to be eligible to participate in this study:

1. Chinese healthy adult males, female subjects (either gender the proportion of not less than 1 / 3).
2. Age: 19 to 45 (including 19, 45) years old.
3. Male body weight ≥ 50kg, female body weight ≥ 45kg, and body mass index within the normal range (weight (kg) / height 2 (m2) = 18-25).
4. Informed consent form is obtained.

Exclusion Criteria:

Subjects will be excluded from entry if any of the criteria listed below are met:

1. Presence or history of any disorder of cardiovascular system, respiratory system, digestive system, urogenital system, endocrine system, allergy / immune system, blood system, nervous / mental system, musculoskeletal system, skin diseases.
2. History of any drug hypersensitivity.
3. Female urine pregnancy test was positive.
4. Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), hepatitis B e antigen (HBeAg), and/or hepatitis C virus (HCV) antibodies.
5. Acute disease state or infection associated with prescription drugs within 1 month before study day 1.
6. Taking any drugs, including over-the-counter drugs and herbal supplements within 7 days before study day 1.
7. History of alcohol abuse (consuming greater than 14 glasses of alcoholic beverages each week, 1 glass is approximately equivalent to: beer 284 mL, wine 125 mL, or distilled spirits [25 mL).
8. History of drug abuse.
9. Smoker or subjects quitting smoking less than 1 month before study day 1.
10. Participating other trials within 1 month before study day 1.
11. Donating blood (> 400 mL) within 1 month before study day 1.
12. During screening, alcohol breath test result > 0.000.
13. Systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg.
14. Heart rate was lower than 45 beats per minute (bpm) and/or higher than 90 bpm during rest.
15. The investigator thought the subjects might not be able to complete the study or comply with the requirements of the study (due to management reasons or other reasons).

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The maximum observed plasma concentration | predose and at 1, 3, 5, 7, 9, 12, 15, 20, 30, 60 and 90 minutes postdose
area under the concentration-time curve | predose and at 1, 3, 5, 7, 9, 12, 15, 20, 30, 60 and 90 minutes postdose
clearance | predose and at 1, 3, 5, 7, 9, 12, 15, 20, 30, 60 and 90 minutes postdose
volume of distribution | predose and at 1, 3, 5, 7, 9, 12, 15, 20, 30, 60 and 90 minutes postdose
terminal half-life | predose and at 1, 3, 5, 7, 9, 12, 15, 20, 30, 60 and 90 minutes postdose
amount excreted in urine | predose and at 1, 3, 5, 7, 9, 12, 15, 20, 30, 60 and 90 minutes postdose
renal clearance | predose and at 1, 3, 5, 7, 9, 12, 15, 20, 30, 60 and 90 minutes postdose
heart rate | predose and at 2, 5, 8, 11, 13, 15, 17, 27 and 42 minutes postdose

CONTACTS AND LOCATIONS:
Overall Officials: Ji Jiang, 88068357, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Peking Union Medical College, Beijing, China